CLINICAL TRIAL: NCT02996799
Title: Efficacy and Safety of Deferred Umbilical Cord Clamping Compared to Umbilical CordMilking in Preterm Infants: A Randomized Clinical Trial
Brief Title: Deferred Cord Clamping Compared to Umbilical Cord Milking in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Heidi Al-Wassia, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 409-16
Record Dates: First submitted 2016-12-03; First posted 2016-12-19 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2021-09

CONDITIONS: PreTerm Birth; Intraventricular Hemorrhage
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferred Cord Clamping (No Intervention): Neonate is held at the level of placenta (level of introitus (vaginal delivery ) and mother's thigh or operating table (C/S) and cord clamping is deferred for 60 seconds.
- Umbilical cord milking (Experimental): Manually stripping 20cm of cord segment toward the umbilicus over a period of 2-3 seconds three times before cord clamping.
  Interventions: Other: Umbilical cord milking

INTERVENTIONS:
Other: Umbilical cord milking — Milking of the umbilical cord at delivery
  Arms: Umbilical cord milking

SUMMARY:
For preterm infants, deferred cord clamping has been shown to improve both short term and long-term neonatal outcomes without an established harm for both the mother and her infant.The interference with resuscitative measures for the neonate or the mother is a risk that continued to hamper the implementation of delayed cord clamping in many centers around the world.For that reason, the evidence now is seeking a time-honored, yet not adopted method of placental transfusion that involves milking of the umbilical cord.

DETAILED DESCRIPTION:
Contrary to delayed cord clamping, milking of the umbilical cord is done at a faster rate and in shorter time.Recent evidence has demonstrated the efficacy and safety of umbilical cord milking for both term and preterm infants.A newer evidence comparing delayed cord clamping to umbilical cord milking in preterm infants demonstrated a higher initial hemoglobin, blood pressure and systemic blood flow in preterm infants allocated to the umbilical cord milking arm.However, concerns have been raised with regard to rapid infusion of large volume of blood in relatively shorter time predisposing to hyperperfusion injury including intraventricular hemorrhage. This is particularly problematic for preterm neonates as they are at higher risk of neurological injury. It has, though, advantage of shorter timeframe allowing for effective resuscitation of preterm neonates to start as soon as possible. Thus, with countering advantages and disadvantages, the practice has not been adopted at most places. The authors planned to conduct a randomized clinical trail to compare the efficacy and safety of umbilical cord milking to deferred cord clamping in preterm infants less than 32 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 32 weeks gestation confirmed by first trimester US

Exclusion Criteria:

* Any proven or suspected congenital or chromosomal abnormalities
* Placenta previa or abruption
* Cord prolapse
* Known Rh sensitization
* Fetal hydrops
* Monochorionic multiples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Intraventricular haemorrhage | twenty eight days
  Any IVH diagnosed by cranial ultrasound

SECONDARY OUTCOMES:
Need for resuscitation | one hour
  Cardiac compression or medications at birth
Apgar score at one minute | one minute after delivery
  Calculated Apgar score at one minute
Apgar score at 5 minutes | 5 minutes after delivery
  Calculated Apgar score at 5 minutes
The need for blood transfusion during hospital stay | one month
  The number of blood transfusions during hospital stay
Venous Hgb | 2 days
  Hgb at birth
Venous hematocrit | 2 days
  Hematocrit at birth
Bilirubin level | 24 hours after birth
  First bilirubin level after birth
Maximum bilirubin level | first week of life
  Highest bilirubin level
Polycythemia | first 48 hours after birth
  If venous hematocrit more than 65%
Respiratory distress syndrome | 48 hours after birth
  The need for surfactant administration
Oxygen dependency | first 28 days after birth and 36 weeks corrected age
  first 28 days after birth and/or 36 weeks corrected age
Need for volume administration | 24 hours after birth
  Need for bolus administration first 24 hours after birth
Use of inotropes | First 24 hours
  Use of any kind of inotropes in the first 24 hours
Necrotizing enterocolitis | one month
  Bell stage II or more
Mortality in hospital | one month
  Death before discharge
Sepsis | one month
  Positive blood culture
Maternal mortality | 2 weeks
  Maternal death after delivery in hospital
Post partum hemorrhage | one day
  Maternal estimated blood loss more than 500 mls in the first 24 hours after birth
Maternal need for blood transfusion | First 48 hours after delivery
  Maternal blood transfusion in the first 48 hours after delivery
Length of third stage | 24 hours
  The time from delivery of the infant until delivery of placenta

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Al-Wassia, MD, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
We are planning to publish all the data that we will collect. If other researchers have specific questions about the data, we are willing to answer and share if needed.
Supporting Information: Study Protocol
Time Frame: Data will be available upon request
Access Criteria: Shared files